CLINICAL TRIAL: NCT04378504
Title: Evaluation of in- Hospital Course of Acute Coronary Syndromes in the Contempory Area
Brief Title: In Hospital Course of Acute Coronary Artery Syndromes
Acronym: HACSA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0271
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Acute Coronary Syndrome; Intensive Care Unit Syndrome
Keywords: Acute coronary syndromes; Intensive care unit; Coronary angiography; In hospital events
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACS: All patients admitted in the ICU for ACS after coronary angiography evaluation between May 2019 and May 2020

SUMMARY:
While international guidelines have indicated that use of a routine invasive strategy was favored for high-risk patients with NSTE-ACS and for all STE- ACS, the lower risk patients successfully reperfused and carrefully selected may perhaps not benefit of this systematic strategy. Evaluation of complications occurring in a contemporary population of ACS may help to evaluate the need of ICU strategy. Coupled with favorable outcomes in many patients, these data may be an opportunity for testing of strategies to refine triage to less costly hospital care units. The investigators thus want to compare, through an observational and prospective study, the event rate of two groups of patients with ACS admitted to ICU . Patients are classified as "high risk" and "low risk" according to specific medical criteria validated in the literature. The study will include all consecutive patients admitted for NSTACS and STACS admitted to the intensive care department of the Montpellier university hospital with the diagnosis of ACS confirmed by coronary angiography.

Our primary goal is to compare the percentage of patients with at least one serious clinical event between the high and low risk groups. A serious event is defined by the occurrence within 7+/-5 days of one of the following criteria: death all causes, serious neurological or hemorrhagic complications, hemodynamic instability and severe heart failure, rhythm or sustained or poorly tolerated conduction disorders requiring therapeutic intervention, painful recurrence requiring new coronary angiography, secondary transfer to intensive care for any reason.

Our hypothesis is that low-risk patients will have very few events and no fatal events and that they could not require intensive care unit admission .

DETAILED DESCRIPTION:
All patients admitted in the ICU Montpellier University center for ACS from May 2019 to May 2020 will be evaluated and classed as low risk patients (groupe LR) or not low risk patients (NLR) after coronary angiography evaluation. High risk criteria will include age >80 years, severe comorbidities, unstable hemodynamic or rhythmic state requiring specific therapeutic intervention, failure of reperfusion or unsatisfactory result of angioplasty, patients with residual coronary lesions requiring further revascularization, left ventricular ejection fraction <40%. Patients who have not received optimal antithrombotic treatment during angioplasty for any reason will also be considered at high risk, as will patients at risk of bleeding due to antecedent or associated pathology or taking a long-term anticoagulant treatment. For the specific case of SCA with ST segment elevation, they will all be included in the group, except for patients who have been successfully reperfused less than 3 hours after the onset of pain or who have an open artery during coronary angiography performed within the first 3 hours.

Our primary endpoint is to compare the percentage of patients with at least one serious clinical event between the high and low risk groups. A serious event is defined by the occurrence within 7+/-5 days of one of the following criteria: death all causes, serious neurological or hemorrhagic complications, hemodynamic instability and severe heart failure, rhythm or sustained or poorly tolerated conduction disorders requiring therapeutic intervention, chest pain recurrence requiring new coronary angiography, any secondary transfer to intensive care for any reason. Secondary endpoints include evaluation of adverse events (all-cause and cardiovascular mortality, unplanned hospitalization for cardiac and non-cardiac causes) at 1 month follow-up in the 2 groups, length of hospitalization of the two groups, calculation of the average number of serious events per patient The low-risk group event rate is estimated at 3 percent without any fatal events. It is estimated at 15 percent in the high risk group.

Assuming a frequency of the event of 3% in the low risk group and 15% in the high risk group, it is necessary to include at least 269 patients, including 196 patients in the high risk group and 73 patients in the low risk group (for a power of 90% and an alpha risk of 5%).

Our hypothesis is that low-risk patients, about 1/3 of ACS admission in ICU, will have very few events and no fatal events and that they don't need intensive care admission

ELIGIBILITY:
Inclusion criteria:

* ACS with or without ST elevation during the inclusion period (May 2019 to May 2020)
* Patients all admitted in ICU after coronary angiography and angioplasty if required

Exclusion criteria:

* Patients not admitted in ICU
* Patients without coronary angiography evaluation
* lack of patient consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in the ICU for ACS after coronary angiography evaluation between May 2019 and May 2020
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
clinical evaluation during hospitalization | 1 day
  all causes of death, serious neurological or hemorrhagic complications, hemodynamic instability and severe heart failure, rhythm or sustained or poorly tolerated conduction disorders requiring therapeutic intervention, chest pain recurrence requiring new coronary angiography, secondary transfer to intensive care for any reason

SECONDARY OUTCOMES:
all-cause and cardiovascular mortality | 1 month
  all-cause and cardiovascular mortality, unplanned hospitalization for cardiac and non-cardiac causes) at 1 month follow-up in the 2 groups, length of hospitalization of the two groups, calculation of the average number of serious events per patient : One month follow up (by phone or medical consultation)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Akodad M, Meunier PA, Padovani C, Cayla G, Zitouni W, Macia JC, Robert P, Steinecker M, Roubille F, Leclercq F. Identification of Low- versus High-Risk Acute Coronary Syndrome for a Selective ECG Monitoring Strategy. J Clin Med. 2023 Jul 11;12(14):4604. doi: 10.3390/jcm12144604. PMID 37510718